CLINICAL TRIAL: NCT02457494
Title: CALVIH: Determination of Kidney Stone Risk Factors in Patients Infected With HIV
Brief Title: Kidney Stone Risk Factors in Patients Infected With HIV
Acronym: CALVIH
Status: Completed | Type: Observational
Sponsor: Corinne Isnard Bagnis (Other)
Responsible Party: Sponsor-Investigator, Corinne Isnard Bagnis, University Professor and Hospital Practitioner, Association pour le Developpement d'Investigations et de Thérapeutiques en Néphrologie
Organization: Association pour le Developpement d'Investigations et de Thérapeutiques en Néphrologie (Other)
Other Study IDs: Al424-986
Record Dates: First submitted 2015-05-22; First posted 2015-05-29 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Nephrolithiasis; HIV
Keywords: CALVIH; Renal stone; HIV1; Renal colic; Atazanavir; Crystalluria; Chronic Kidney Disease; Calcium Oxalate
MeSH Terms: conditions — Nephrolithiasis; Renal Colic; Crystalluria; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to define the cause of renal stones and the risk pattern for recurrence of renal stones episodes (any kind of stones) in HIV1 patients.

DETAILED DESCRIPTION:
This study aims at defining the cause of renal stones and the risk pattern for recurrence of renal stones episodes (any kind of stones) in HIV1 patients.

Primary Objective :

* Finding the cause of renal stone in HIV patients defined as stone composition if stone is available or more probable pathophysiological mechanism
* Risk profile for stone recurrences estimated on risk indices in HIV1 patients

Secondary Objective(s)

* Identify prevalence of recurrences and describe co-morbidities associated with stone disease
* Describe urological management for renal stones in HIV patients
* Describe the causes of drug induced renal stones

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female HIV1 infected patients willing to participate in the study
* Having experienced a renal stone episode within the past six months or living with a renal stone
* Able to understand the protocol
* Giving oral consent

Exclusion Criteria:

* CT scan impossible
* Follow up impossible over 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female HIV1 infected patients having experienced a renal stone episode within the past six months or living with a renal stone
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-05; Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of the cause of the renal stone | at 6 months
  Qualitative assessment of the cause of the renal stone based on different biological and clinical parameters (biochemical analysis of urines, cristalluria, low dose renal CT, patient history, family history…)
Risk profile for recurrence of renal stone | at 12 months
  Risk profile for recurrence of renal stone estimated based on plasma and urinary parameters, nutritional profile and drug exposure

SECONDARY OUTCOMES:
Follow up outcome of HIV patients over one year to identify prevalence of recurrences and describe co-morbidities associated with stone disease | up to 12 months
Urological management for renal stones in HIV patients | up to 12 months
Causes of drug induced renal stones | up to 12 months
Number of stone recurrences | at 6 months
Number of stone recurrences | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: corinne i bagnis, Principal Investigator — Groupe Hospitalier Pitie Salpetriere et Chaire de Recherche en Education Therapeutique
Locations (1):
- Corinne Isnard Bagnis, Paris, France

REFERENCES:
- [Result] Abgrall S, Rachas A, Tourret J, Isnard-Bagnis C, Billaud E, Tattevin P, Costagliola D, Guiguet M, Durieux P; French Hospital Database on HIV. A multifaceted intervention designed to improve medical management of moderate to advanced chronic kidney disease in HIV-infected patients: a cluster randomized trial. Clin Infect Dis. 2015 Aug 1;61(3):375-84. doi: 10.1093/cid/civ310. Epub 2015 Apr 22. PMID 25904366
- [Result] Tourret J, Deray G, Isnard-Bagnis C. Tenofovir effect on the kidneys of HIV-infected patients: a double-edged sword? J Am Soc Nephrol. 2013 Oct;24(10):1519-27. doi: 10.1681/ASN.2012080857. Epub 2013 Sep 19. PMID 24052632
- [Result] Bige N, Lanternier F, Viard JP, Kamgang P, Daugas E, Elie C, Jidar K, Walker-Combrouze F, Peraldi MN, Isnard-Bagnis C, Servais A, Lortholary O, Noel LH, Bollee G. Presentation of HIV-associated nephropathy and outcome in HAART-treated patients. Nephrol Dial Transplant. 2012 Mar;27(3):1114-21. doi: 10.1093/ndt/gfr376. Epub 2011 Jul 10. PMID 21745806
- [Result] Tourret J, Tostivint I, Deray G, Isnard-Bagnis C. [Kidney diseases in HIV-infected patients]. Nephrol Ther. 2009 Nov;5(6):576-91. doi: 10.1016/j.nephro.2009.02.007. Epub 2009 Apr 16. French. PMID 19375399